CLINICAL TRIAL: NCT04696211
Title: A Music-with-movement Exercise Program for Community-dwelling Older Adults Suffering From Chronic Pain: a Pilot Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MMEP
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Chronic Pain; Elderly; Music-with-movement Exercise; Pain Management
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The music-with-movement exercise program (MMEP) is an 8-week program. In the first 4 weeks a center-based program will be offered in the District Elderly Centers, and from week 1 to week 8 home-based and digital-based activities will be delivered via a WhatsApp group.
  Interventions: Other: Music-with-movement exercise
- Control group (No Intervention): The participants in the control group will continue to receive their usual care and receive a one-page pain management pamphlet.

INTERVENTIONS:
Other: Music-with-movement exercise — A music-with-movement exercise programme to reduce chronic pain in older adults.
  Arms: Experimental group

SUMMARY:
Background: The high prevalence of chronic pain in community-dwelling older adults requires attention from nurses. The aim of the present study is to use a music-with-movement exercise program to improve the pain situations of older adults with chronic pain.

Aims and objectives:

The aim of this study is to implement a music-with-movement exercise program (MMEP) for older adults suffering from chronic pain.

The objectives of this study are:

* To evaluate the effects of a music-with-movement exercise program on improving the pain intensity, pain self-efficacy, mood, and quality of life of the older adults with chronic pain
* To observe the participants' level of adherence to the music-with-movement exercise by using an exercise logbook and measurements of heart rate

Anticipated outcomes: This study will be a pilot randomized controlled trial. An 8-week music-with-movement exercise program will be used as the intervention for older adults with chronic pain in District Elderly Centers in Hong Kong. It will consist of four sessions of center-based, face-to-face activities and four weeks home-based and digital-based activities delivered through a WhatsApp group. A music therapist, in consultation with the physiotherapist, will lead the center-based activities. Each center-based session will consist of 30 minutes of music-with-movement exercise and 10 minutes of instruction on pain knowledge and pain management. Each participant will receive an exercise logbook to practice and record the frequency of their engagement in the music-with-movement exercise at home. They will receive WhatsApp reminders to remind them to continue the home-based sessions. Outcome measures include pain intensity, pain self-efficacy, mood, heart rate and physical activity intensity, and quality of life. Data will be collected before and after the intervention. Participants need to complete the exercise logbook to record their adherence to the intervention. The findings of this study will provide clinical implications for nurses to integrate music with movement exercise to manage pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or above
* Can understand Cantonese
* Have a history of non-cancer pain in the past 3 months
* Have a pain score of at least 2 as measured by the Numeric Rating Scale (on an 11-point numeric scale)
* Able to take part in an exercise and stretching program
* Owns a smartphone and can access the Internet

Exclusion Criteria:

* Have severe visual and/or auditory deficits
* Have a serious organic disease or malignant tumor
* Have a mental disorder diagnosed by neurologists or psychiatrists
* Had surgical treatments in the past two months
* Experienced drug addiction

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, Week 8
  Changes from baseline to Week 8 in pain intensity using the Chinese version of Brief Pain Inventory (BPI-C)

SECONDARY OUTCOMES:
Pain self-efficacy | Baseline, Week 8
  Changes from baseline to Week 8 in pain self-efficacy using the Chinese version of Pain Self-efficacy Questionnaire
Loneliness | Baseline, Week 8
  Changes from baseline to Week 8 in loneliness using the Chinese version of De Jong Gierveld Loneliness Scale
Depression | Baseline, Week 8
  Changes from baseline to Week 8 in depression using the Chinese version of Geriatric Depression Scale
Satisfaction and acceptability | Week 8
  Questions designed by the research team to collect the participants' satisfaction and acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Mimi MY Tse, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: Undecided